CLINICAL TRIAL: NCT04361825
Title: Phase Ⅱ, Single-arm Study of Durvalumab(MEDI4736) and AZD6738 Combination Therapy in Relapsed Small Cell Lung Cancer Subjects [SUKSES-N4]
Brief Title: Durvalumab(MEDI4736) and AZD6738 Combination Therapy in Relapsed Small Cell Lung Cancer Subjects
Acronym: SUKSES-N4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Se-Hoon Lee (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Se-Hoon Lee, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02-103
Record Dates: First submitted 2020-04-12; First posted 2020-04-24 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; ceralasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab(MEDI4736) and AZD6738 combination (Experimental)
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500mg via IV administered for every 4weeks(fixed dosing for subjects > 30 kg body weight) in Day 1 of each cycle and AZD 6738 240mg bid per os administered in each cycle days 1 and 7. One cycle is consisted of 28 days.
  Other Names: AZD6738

SUMMARY:
This study is a single arm, multi-center phase II study of durvalumab and AZD6738 combination therapy in subjects with relapsed small cell lung cancer (SCLC) as a second or third line chemotherapy.

DETAILED DESCRIPTION:
Subjects will receive durvalumab and AZD6738 combination therapy. The arm is composed of 45 subjects.

Durvalumab 1500mg via IV administered for every 4weeks(fixed dosing for subjects > 30 kg body weight) in Day 1 of each cycle and AZD 6738 240mg bid per os administered in each cycle days 15 and 28. One cycle is consisted of 28 days.

Tumour evaluation using CT or MRI, RECIST 1.1, CEA, NSE and LDH will be conducted at screening (within 28days prior to first dose of Cycle1 Day1) and every 8weeks(±1week) for the first 56weeks relative to the start of combination therapy(Cycle1 Day1), and thereafter every 12weeks(±1week) until objective disease progression.

Study treatment will be continued until objective disease progression (unless other criteria for treatment discontinuation are met). Subjects may continue durvalumab and AZD6738 beyond progression(according to RECIST 1.1), at the discretion of the investigator if they are clinically benefiting from the treatment and they do not meet any other discontinuation criteria.

If a subjects discontinues study treatment prior to disease progression, they should continue to be assessed using RECIST 1.1 until disease progression and then followed up for survival.

Assessments for survival should be made every 3months following objective disease progression. The details of first and subsequent therapies for cancer, after discontinuation of durvalumab and AZD6738 treatment, will be collected.

The imaging modalities used for RECIST 1.1 assessment will be CT or MRI scans of chest, abdomen and pelvis. And CEA, NSE and LDH tests are also used for the evaluation. RECIST 1.1 scans will be analysed by the investigator on site.

Subjects may also be requested to provide tumour samples from the primary or metastatic tumours on progression to understand resistance mechanisms. Sample provision is optional and depend on the subject's will.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Subjects must be ≥ 18years of age.
3. Body weight > 30kg
4. Small cell lung cancer that has progressed during or after first-line therapy.

   1. The 1st line regimen must have contained platinum based regimen and must have documented radiological and/or clinical progression on treatment. The subjects must not exposed to the prior immunotherapy which could have been received separately, in combination, or in sequence with platinum-doublet chemotherapy.
   2. Refractory to first-line chemotherapy or relapse within 6months since the last dose of first-line chemotherapy
   3. If the subject correspond to sensitive relapse(relapse more than 6months since the last dose of first-line chemotherapy), (s)he should get second-line treatment prior to study entry.
5. Subjects are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
6. ECOG performance status 0-1
7. Subjects must have a life expectancy ≥ 3months from proposed first dose date.
8. Subjects must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   1. Haemoglobin ≥ 9.0g/dL
   2. White blood cells(WBC) ≥ 3 x 109/L
   3. Platelet count ≥ 100 x 109/L
   4. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   5. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   6. Aspartate aminotransferase(AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase(ALT) (Serum Glutamic Pyruvate Transaminase(SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN
   7. Subjects must have serum creatinine (CR)≤1.5 times the normal upper limit of the study institution or creatinine clearance estimated using the Cockcroft-Gault equation of ≥ 45 mL/min
9. At least one measurable lesion that can be accurately assessed at baseline by imaging or physical examination at baseline and is suitable for repeated assessment.
10. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test test at screening and confirmed prior to treatment on Day 1 of every cycle Postmenopausal is defined as:

    1. Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    2. Luteinizing hormone(LH) and Follicle stimulating hormone(FSH) levels in the post menopausal range for women under 50
    3. Radiation-induced oophorectomy with last menses >1 year ago
    4. Chemotherapy-induced menopause with >1 year interval since last menses surgical sterilisation(bilateral oophorectomy or hysterectomy
11. Male Subjects and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination for acceptable methods, throughout the period of taking study treatment and for 6months after last dose of investigational product(s) to prevent pregnancy in a partner.
12. Provision of informed consent for genetic research. If a subject declines to participate in the genetic research, there will be no penalty or loss of benefit to the subject.

Exclusion Criteria:

1. Previous enrolment in the present study.
2. More than two prior chemotherapy regimen for the treatment of small cell lung cancer(However, immunotherapy is not counted the prior chemotherapy regimen.)
3. Subjects with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for > 2years.
4. Treatment with any investigational product during the last 14days before the enrollment (or a longer period depending on the defined characteristics of the agents used).
5. Subjects receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The subject can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4weeks prior to treatment.
6. Rceiving, or having received, concomitant medications, herbal supplements and/or foods that significantly modulate cytochrome P450 3A4(CYP3A4) or P-glycoprotein(P-gp) activity(washout periods of 2weeks, but 3weeks for St. John's Wort). Note these include common azole antifungals, macrolide antibiotics and other medications.
7. Prior exposure to an ATR inhibitor.
8. Refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection, with clinically significant sequelae that would preclude adequate absorption of AZD6738
9. Current or prior use of immunosuppressive medication within 14days before the first dose of durvalumab. The following are exceptions to this criterion:

   1. Intranasal, inhaled, topical steroids, or local steroid injections(eg, intra-articular injection)
   2. Systemic corticosteroids at physiologic doses not to exceed 10mg/day of prednisone or its equivalent
   3. Steroids as premedication for hypersensitivity reactions(eg, CT scan premedication)
10. Receipt of live attenuated vaccine within 30days prior to the first dose of investigational product. Note: Subjects, if enrolled, should not receive live vaccine whilst receiving investigational product and up to 180days after the last dose of investigational product.
11. Any unresolved toxicity NCI CTCAE grade≥2 from previous anticancer therapy with the exception of alopecia, vitilgo, and the laboratory values defined in the inclusion criteria(CTCAE 5.0)

    1. Subjects with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    2. Subjects with irreversible toxicity not reasonably expected tobe exacerabated by treatment with durvalumab may be included only after consultation with with the Study Physician.
12. Intestinal obstruction or CTCAE 5.0 grade 3 or grade 4 upper GI bleeding within 4weeks before the enrollment.
13. Haematuria: +++ on microscopy or dipstick
14. INR ≥ 1.5 or other evidence of impaired hepatic synthesis function
15. Subject has any of the following cardiac criteria:

    1. Mean QT interval corrected for heart rate(QTc) ≥ 470ms calculated from 3 electrocardiograms(ECGs) using Fridericia's correction.
    2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block, second degree heart heart block, first degree heart block.
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40years of age or any concomitant medication known to prolong the QT interval.
    4. Uncontrolled hypertension-blood pressure (BP) ≥ 150/95mmHg despite medical therapy.
    5. Unstable atrial fibrillation or unstable cardiac arrhythmia with a ventricular rate > 100bpm on an ECG at rest.
    6. Symptomatic heart failure - New York Heart Association Grade II to Grade IV.
    7. Prior or current cardiomyopathy.
    8. Severe valvular heart disease.
    9. Uncontrolled angina (Canadian Cardiovascular Society Grade II to Grade IV despite medical therapy) or acute coronary syndrome within 6months prior to screening.
    10. Subjects at risk of brain perfusion problems (e.g., carotid stenosis hypotension, including a fall in blood pressure of > 20mm Hg)
16. Female subjects who are pregnant or breast-feeding or child-bearing or male or female subjects of of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
17. Any evidence of severe or uncontrolled intercurrent illness, including but limited to, ongoing or active infection, symptomatic conjestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent.
18. History of allogenic organ transplantation.
19. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B(known positive HBV surface antigen(HBsAg) result), Hepatitis C, or human immunodeficiency virus(positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the antibody[anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C(HCV) antibody are eligible only if polymerage chain reaction is negative for HCV RNA.
20. Known hypersensitivity to any of study drug or any of the study drug excipients.
21. Known central nervous system(CNS) disease other than neurologically stable,treated brain metastases - defined as metastasis having no evidence of progression or haemorrhage for at least 2weeks after treatment.
22. Major surgical procedures ≤ 28days of beginning study treatment, or minor surgical procedures≤ 7days
23. History of active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis [with the exception of diverticulosis], systemic lupus erythematosis, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).

The following are exceptions to this criterion:

1. Subjects with vitiligo or alopecia
2. Subjects with hypothyroidism(e.g., following Hashimoto syndrome) stable on hormone replacement
3. Any chronic skin condition that dose not require systemic therapy
4. Subjects without active disease in the last 5 years may be included but only after consultation with the study physician
5. Subjects with cardiac disease controlled by diet alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Efficacy of durvalumab and AZD6738 combination therapy in subjects with relapsed SCLC subjects as 2nd or 3rd line therapy: Objective response rate(ORR) | Up to 30 months
  Objective response rate(ORR) by RECIST 1.1

SECONDARY OUTCOMES:
Duration of response | Up to 30 months
  Duration of response (DOR) is the time from the date of the first dose of study treatment to the date of RECIST progression or death from any cause, whichever occurs first.
Disease control rate | 8 weaks
  Disease control rate (DCR) is the number of patients having a CR or PR or stable disease via RECIST divided by the number of patients in the full analysis set.
Overall survival(OS) | Up to 30 months
  Overall survival (OS) is the time from the date of the first dose of study treatment to the date of death from any cause.
progression-free survival(PFS) | Up to 30 months
  Progression-free survival (PFS) is the time from the date of first dose of study treatment to the date of RECIST progression or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hoon Lee, M.D,Ph.D., Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No